CLINICAL TRIAL: NCT06800352
Title: Investigation of the Effect of Olive Oil and Centaury Oil in the Management of Diaper Dermatitis
Brief Title: The Effect of Olive Oil and Centaury Oil on Rash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, HASRET YAĞMUR SEVİNÇ AKIN, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HRU-VSYO-HYSA-2024/139
Record Dates: First submitted 2025-01-03; First posted 2025-01-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diaper Dermatitis
Keywords: olive oil; centaury oil; diaper dermatitis
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Intervention Model Description: Block randomisation method will be used in this study. Using the online programme (http://www.randomizer.org), a random list of sets assigning infants to groups will be created. The infants who will constitute the sample of the study will be divided into 20 sets with 3 people in each set and sets will be formed by assigning numbers from 1 to 3 to each set. When the sets are obtained, the numbers from 1 to 3 will be written on small papers and group assignments will be made by lot method. In this way, the number of babies included in the groups and the probability of each baby to be included in the study groups will be equalised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Oil Application (Experimental): The degree of diaper dermatitis will be evaluated before and after the procedure (72 hours after the first procedure) using the 'Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants'. After cleaning the perineum as described to the mothers, they will be asked to apply olive oil to the perineum four times a day, 1 cc each time.
  Interventions: Other: Control
- Centaury Oil Application (Experimental): The degree of diaper dermatitis of the infants will be evaluated before and after the procedure (72 hours after the first procedure) using the 'Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants'. After cleaning the perineum as described to the mothers, they will be asked to apply centaury oil to the perineum four times a day, 1 cc each time.
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — The degree of diaper dermatitis of the babies will be evaluated before and after the procedure (72 hours after the first procedure) by using the 'Uncomplicated Diaper Dermatitis Severity Rating Scale in Babies (UNDDCS)'. Mothers will be asked to diaper their babies with cotton wool soaked with clear water.

SUMMARY:
Diaper dermatitis is a preventable health problem. No study evaluating the efficacy of centaury oil in diaper dermatitis was found in the literature. This study will be conducted to investigate the effect of olive oil and centaury oil in the management of diaper dermatitis.

DETAILED DESCRIPTION:
Diaper dermatitis is estimated to have an incidence of between 7% and 35%, although the prevalence cannot be determined precisely because it is not usually seen as a disease by parents and most patients are treated at home. Prevention of diaper dermatitis should be the main approach in treatment and care. Once it occurs, the aim of treatment is to accelerate the healing of the damaged area and prevent its spread. In the prevention and treatment of diaper dermatitis, practices such as ventilating the baby's diaper, changing the diaper frequently, keeping the area dry, cleaning with appropriate methods, using barrier creams and not tying the diaper tightly have been reported to be beneficial.

In the literature, studies using methods such as water, herbal cream (chamomile cream, calendula cream, aloe vera cream), barrier cream (zinc oxide) and herbal mixture (honey, beeswax, olive oil) were found in the treatment of infants with mild to moderate diaper dermatitis. It has been stated that the rates of diaper dermatitis will continue to increase if parents are not given adequate information about appropriate care and which products are beneficial or even harmful. In conclusion, diaper dermatitis is a preventable health problem. No study evaluating the efficacy of olive oil and centaury oil in diaper dermatitis was found in the literature. This study will be conducted to examine the effect of olive oil and centaury oil in the management of diaper dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* The baby has mild diaper dermatitis according to the diaper dermatitis severity rating scale
* The baby receives antibiotic treatment
* The baby gets additional food
* The baby is between 6-18 months

Exclusion Criteria:

* Infants with moderate or severe diaper dermatitis according to the diaper dermatitis severity rating scale
* Babies with open wounds on the perineum,
* Babies with any skin disease
* Babies who use barrier creams or special oils in routine care

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Outcome Measures | 1 year
  The outcome measures for the sociodemographic data of the study will be collected by using the 'Introductory Information Form', which includes questions about the infant's identifying characteristics such as gender, age, height, weight and diaper care.
  The other outcome measure to be used in the study is the 'Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants' which will be used to rate the severity of diaper dermatitis in infants.
  Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants: The lowest score that can be obtained from the scale consisting of a total of four items is zero and the highest score is six. The minimum and maximum scores that can be obtained from each item are 0-3 points for the severity of erythema or irritation item, 0-1 point for the degree of diaper dermatitis item, 0-1 point for the papules and pustules item and 0-1 point for the open skin item. As the score on the scale increases, the degree of diaper dermatitis also increases

CONTACTS AND LOCATIONS:
Overall Officials: H YAĞMUR SEVİNÇ AKIN, Assistant Professor, Study Director — Harran University; MAKSUDE YILDIRIM, Assistant Professor, Principal Investigator — Adiyaman University; BARIŞ AKIN, Specialist nurse, Principal Investigator — Mardin Training and Research Hospital; NESRİN ŞEN CELASİN, Assoc. Professor, Principal Investigator — Celal Bayar University; ZÜLEYHA GÜRDAP, RESEARCH ASSISTANT, Principal Investigator — Inonu University
Locations (1):
- Mardin Training and Research Hospital, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No